CLINICAL TRIAL: NCT07321483
Title: Evaluation of the Therapeutic Efficacy of Reflex Therapy Using Dry Needling in Patients With Functional Temporomandibular Pain Syndrome: A Prospective, Randomized, Controlled Pilot Study.
Brief Title: Reflex Therapy of Temporomandibular Dysfunctions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Petr Konecny, Associate Professor, Head of the Institute of Clinical Rehabilitation, Palacký University Olomouc, Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGA_FZV_2025_015
Record Dates: First submitted 2025-11-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Dysfunction; Myofascial Pain Syndrome; Orofacial Pain; Musculoskeletal Disorders
Keywords: headache; temporomandibular disorders; dry needling; rehabilitation therapy; pain; quality of life; temporomandibular disorders; dry needling; rehabilitation therapy; pain; quality of life
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes; Facial Pain; Musculoskeletal Diseases; Headache; Pain | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: intervention with Dry Needling and Standard Rehabilitation) (Experimental): Participants in this group will receive standard outpatient rehabilitation therapy combined with Intervention: one dry needling intervention targeting trigger points in the masseter and temporalis muscles during the first treatment session. The rehabilitation program will include mobilization, soft tissue techniques, and targeted kinesiotherapy. Each participant will undergo ten outpatient rehabilitation sessions over five weeks (two sessions per week).
  Interventions: Procedure: Dry needling; Procedure: Standard rehabilitation
- Control Group - Standard Rehabilitation (Active Comparator): Participants in this group will receive the same standard outpatient rehabilitation program as the experimental group, excluding the dry needling procedure. The therapy will include mobilization, soft tissue relaxation techniques, and specific exercises focused on improving temporomandibular joint mobility and reducing muscle tension
  Interventions: Procedure: Standard rehabilitation

INTERVENTIONS:
Procedure: Dry needling — One dry needling intervention targeting trigger points in the masseter and temporalis muscles during the first treatment session
  Other Names: reflex injection therapy of Trigger Point
  Arms: Experimental Group: intervention with Dry Needling and Standard Rehabilitation)
Procedure: Standard rehabilitation — The therapy will include mobilization, soft tissue relaxation techniques, and specific exercises focused on improving temporomandibular joint mobility and reducing muscle tension.
  Other Names: Standard Physical Rehabilitation Program

SUMMARY:
This study aims to evaluate the effectiveness of dry needling in patients with functional temporomandibular pain syndrome by comparing standard rehabilitation therapy alone with therapy combined with dry needling to reduce pain, improve jaw function and enhance quality of life.

DETAILED DESCRIPTION:
This prospective, randomized, controlled pilot study aims to evaluate the therapeutic effects of dry needling in patients with functional temporomandibular pain syndrome. A total of 100 participants will be randomly assigned to two groups: an experimental group receiving standard rehabilitation combined with dry needling therapy, and a control group undergoing standard rehabilitation only. The intervention program will consist of ten outpatient rehabilitation sessions conducted over five weeks.

Outcome measures will include pain intensity (Visual Analogue Scale, VAS), temporomandibular joint range of motion, presence of joint sound phenomena, and quality of life assessed using the World Health Organization Quality of Life - BREF questionnaire (WHOQOL-BREF questionnaire). Measurements will be collected at baseline, immediately after the first therapy session, and upon completion of the treatment cycle.

Descriptive statistics will be used for data analysis. The Shapiro-Wilk test will assess data normality. Between-group differences will be analyzed using parametric (t-test) or nonparametric (Mann-Whitney, Wilcoxon) tests, depending on data distribution. Correlation analyses will be performed using Pearson's or Spearman's correlation coefficients. Statistical significance will be set at p < 0.05.

All statistical analyses will be conducted using IBM SPSS Statistics for Windows, version 29.0 (Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with functional temporomandibular pain syndrome without structural temporomandibular joint damage.
* Aged ≥18 years.
* Stable health condition suitable for outpatient rehabilitation.
* Willingness to participate and ability to follow the therapeutic protocol.

Exclusion Criteria:

* Presence of degenerative, post-traumatic, or inflammatory changes in the temporomandibular joint.
* Cognitive or psychiatric disorders limiting cooperation.
* Lack of informed consent or non-compliance during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
1. Pain Intensity using the Visual Analogue Scale (VAS). | Baseline (pre-intervention) Immediately after the first therapy session At completion of the treatment program (after 10 therapy sessions).
  * Description: Evaluation of subjective pain intensity in the temporomandibular region assessed using the Visual Analogue Scale (VAS), a continuous scale ranging from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain. Higher scores indicate worse pain intensity.
  * Measurement Type: Continuous (0-10 scale).

SECONDARY OUTCOMES:
Temporomandibular Joint (TMJ) Range of Motion, Joint Sound Phenomena and Quality of Life (WHOQOL-BREF) | Baseline (pre-intervention) Immediately after the first therapy session At completion of the treatment program (after 10 therapy sessions)
  * Description: Measurement of maximal mouth opening and mandibular movement range using a caliper to assess functional improvement of the TMJ.
  * Measurement Type: Continuous (millimeters). and
  * Description: Clinical assessment of the presence or absence of joint sounds (clicking, popping, or crepitation) during mandibular movement as an indicator of TMJ functional stability.
  * Measurement Type: Categorical (present/absent). and
  * Description: Evaluation of overall quality of life using the WHOQOL-BREF questionnaire, which assesses physical, psychological, social, and environmental domains.
  * Measurement Type: Continuous (score-based)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Palacký University Olomouc, Czech Republic, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy and institutional data protection policies

REFERENCES:
- [Result] Quilghini C, Lefflot J, Buchholtz K. The effectiveness of physiotherapy for chronic headaches in patients with temporomandibular disorders: a systematic review. Front Rehabil Sci. 2025 Sep 23;6:1647927. doi: 10.3389/fresc.2025.1647927. eCollection 2025. PMID 41064810
- [Result] Armijo-Olivo S, Pitance L, Singh V, Neto F, Thie N, Michelotti A. Effectiveness of Manual Therapy and Therapeutic Exercise for Temporomandibular Disorders: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jan;96(1):9-25. doi: 10.2522/ptj.20140548. Epub 2015 Aug 20. PMID 26294683
- [Result] Konečný P, Havlíčková J, Elfmark M, Tvrdý P, Hanáková D, Jureček M. Effects of Rehabilitation in Patients with Temporomandibular Joint Disorders. Rehabil. Fyz. Lek. (2007) 14: 95-100.